CLINICAL TRIAL: NCT01181453
Title: A Prospective, Multicenter, Randomized, Single-Blind, Phase III, Clinical Investigation of Dermagraft(R) in Patients With Plantar Diabetic Foot Ulcers
Brief Title: Pivotal Trial of Dermagraft(R) to Treat Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABH-DG-04-07-0798
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic foot ulcer; Randomized trial; Clinical trial; Dermagraft; Standard care
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

ARMS (2):
- Dermagraft(R) (Experimental): Weekly application of Dermagraft(R) with standard care
  Interventions: Device: Dermagraft
- Standard care only (Other): Weekly application of standard care
  Interventions: Other: Comparator

INTERVENTIONS:
Device: Dermagraft — Weekly application of Dermagraft(R) with standard care
  Other Names: human fibroblast derived dermal substitute
  Arms: Dermagraft(R)
Other: Comparator — Weekly application of standard care
  Other Names: standard of care, off-loading, surgical debridement, wet-to-moist dressing
  Arms: Standard care only

SUMMARY:
This study randomly assigns patients with diabetic foot ulcers to receive standard therapy (surgical debridement, saline-moistened gauze and offloading) alone or standard therapy plus Dermagraft(R). Dermagraft is a device containing live human fibroblasts grown on an absorbable Vicryl mesh. Patients are seen weekly until they heal or the 12-week treatment period is complete.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient has type I or II diabetes.
* Foot ulcer has been present for a minimum of 2 weeks under the current investigator's care.
* Foot ulcer is on the plantar surface of the forefoot or heel.
* Ulcer size is >/=1.0 cm2 at Day 0 (day of randomization).
* Ulcer extends through the dermis and into subcutaneous tissue but without exposure of muscle, tendon, bone, or joint capsule.
* Ulcer is free of necrotic debris, exhibits no signs of clinical infection, and appears to be made up of healthy vascularized tissue.
* Patient's Ankle-Arm Index by Doppler is >/=0.7.
* Patient has adequate circulation to the foot as evidenced by a palpable pulse.
* Female patients of child bearing potential must not be pregnant and must use accepted means of birth control.
* Patient and caregiver are willing to participate in the clinical study and can comply with the follow-up regimen.
* Patient or his/her legal representative has read and signed the Institutional Review Board (IRB) approved Informed Consent form before treatment.
* Patient's study ulcer has been present (open) for at least 6 weeks at the time of the Screening visit.

Exclusion Criteria:

* There is clinical evidence of gangrene on any part of the affected foot.
* The study ulcer is over a Charcot deformity.
* The study ulcer is due to a nondiabetic etiology.
* The ulcer has tunnels or sinus tracts that cannot be completely debrided.
* The ulcer is >20 cm2 (longest dimension cannot be greater than 5 cm).
* The ulcer has increased or decreased in size by 50% or more during the screening period.
* Presence of medical condition(s) that in the Investigator's opinion makes the patient an inappropriate candidate for this study.
* Presence of a malignant disease not in remission for 5 years or more.
* Evidence of severe malnutrition, based on a serum albumin level <2.0.
* Presence of patient having known alcohol or drug abuse.
* A random blood sugar reading >/=450 mg/dL.
* Presence of urine ketones that are noted to be "Small, Moderate, or Large".
* Presence of a nonstudy ulcer on the study foot within 7.0 cm of the study ulcer at Day 0.
* Use of oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents, Coumadin or heparin during the study.
* A history of bleeding disorder.
* Presence of Acquired Immunodeficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV).
* Participation in another study involving treatment with an investigational product within the previous 30 days.
* Elective osseous procedures to the study foot within 30 days prior to the Screening visit.
* Previous treatment with Dermagraft®.
* Presence in study ulcer of cellulitis, osteomyelitis or other clinical evidence of infection.
* Presence of condition(s) that seriously compromise the patient's ability to complete this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 1998-12; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Complete wound closure | 12 weeks

SECONDARY OUTCOMES:
Time to reach complete wound closure | 12 weeks
Percent of wound closure by study end | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William A Marston, MD, Principal Investigator — University of North Carolina School of Medicine, Chapel Hill, NC
Locations (1):
- University of North Carolina School of Medicine, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Marston WA, Hanft J, Norwood P, Pollak R; Dermagraft Diabetic Foot Ulcer Study Group. The efficacy and safety of Dermagraft in improving the healing of chronic diabetic foot ulcers: results of a prospective randomized trial. Diabetes Care. 2003 Jun;26(6):1701-5. doi: 10.2337/diacare.26.6.1701. PMID 12766097